CLINICAL TRIAL: NCT04860297
Title: A Phase 3b, Open-Label, Safety and Immunogenicity Study of SARS-CoV-2 mRNA-1273 Vaccine in Adult Solid Organ Transplant Recipients and Healthy Controls
Brief Title: A Study to Evaluate Safety and Immunogenicity of mRNA-1273 Vaccine to Prevent COVID-19 in Adult Organ Transplant Recipients and in Healthy Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-1273-P304
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: This is an open-label, single intervention study; there is no randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mRNA-1273 (Experimental): Part A: All participants (healthy participants and SOT participants) who were unvaccinated prior to enrollment will receive 2 intramuscular (IM) injections of 100 microgram (µg) mRNA-1273 on Day 1 and Day 29.
  All SOT participants who were unvaccinated prior to enrollment will be offered the opportunity to receive a third primary dose of mRNA-1273 at Day 85 as per the emergency use authorization (EUA) Fact Sheet available at the time of protocol finalization.
  SOT participants who were previously vaccinated with 2 doses of Moderna COVID-19 vaccine under the EUA prior to enrollment will receive Dose 3 on Day 1.
  Part B: All eligible participants from Part A will be offered to receive a 100 µg booster dose of mRNA-1273 who are at least 4 months from the last dose. SOT recipients who completed primary COVID-19 vaccination series under EUA (outside of the mRNA-1273-P304 study) will receive a 100 µg booster dose on booster dose Day 1.
  Interventions: Biological: mRNA-1273

INTERVENTIONS:
Biological: mRNA-1273 — Sterile liquid for injection

SUMMARY:
This is an open-label study to evaluate the safety, reactogenicity, and immunogenicity of mRNA-1273 Severe Acute Respiratory Syndrome coronavirus (SARS-CoV-2) vaccine in adults with a kidney or liver solid organ transplant (SOT) and in healthy adult participants. The primary goal of the study is to evaluate the safety of mRNA-1273 and the serum antibody (Ab) responses obtained 28 days after the last dose of mRNA-1273.

ELIGIBILITY:
Transplant Recipients

Key Inclusion Criteria for Part A:

* Is either a kidney or a liver transplant recipient who is at least 90 days after transplantation at the time of consent, and is either unvaccinated or previously vaccinated with 2 doses of Moderna COVID-19 vaccine who is at least 1 month after the second dose at the time of consent. Participants who received the 2 doses of Moderna COVID-19 vaccine before transplant are not eligible.
* Understands, agrees, and is able to comply with the study procedures and provides written informed consent.
* Received chronic immunosuppressive therapy for the prevention of allograft rejection for a minimum of 90 days before signing consent, including but not limited to: glucocorticoids (such as, prednisolone), immunophilin binding agents (such as, calcineurin inhibitors, mTOR inhibitors), or inhibitors of de novo nucleotide synthesis (such as, mycophenolic acid, mizoribine, leflunomide, azathioprine).
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection, agreement to continue adequate contraception or abstinence through 3 months following the second dose (Day 29) for those receiving 2-dose regimen and, through 3 months following the third dose (Day 85) for those receiving 3-dose regimen, and through 3 months following the third dose (Day 1) for those previously vaccinated SOT participants, and not currently breastfeeding.
* Is medically stable, according to investigator's judgment, during the 3 months before signing consent.

Key Exclusion Criteria for Part A:

* Has prior or planned administration of a coronavirus vaccine (for example, SARS-CoV-2 [for unvaccinated participants only], SARS-CoV, or MERS [Middle East Respiratory Syndrome] -CoV vaccine).
* Has current treatment with investigational agents for either prophylaxis against COVID-19 (for unvaccinated participants only) or treatment of COVID-19 (such as, anti-SARS-CoV-2 monoclonal antibodies).
* A history of more than one solid organ transplanted (such as, kidney and pancreas). A history of previous kidney or liver transplant is acceptable.
* Has received therapies that have depleting properties on T cells, B cells, and plasma cells (examples of depletional therapies include, but are not limited to, antithymocyte globulin [ATG], monoclonal antibodies, and proteosome inhibitors) within the last 3 months prior to enrollment.
* A history of biopsy-proven T-cell- or Ab-mediated rejection within 3 months of informed consent, or suspected active or chronic rejection according to the investigator's judgment.
* Has a known close contact with anyone with laboratory confirmed SARS-CoV-2 infection within 2 weeks to vaccine administration or known history of SARS-CoV-2 infection or positive SARS-CoV-2 test.
* Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation or that could interfere with safety assessments or interpretation of results according to the investigator's judgment.
* Has a history of clinically relevant donor-specific Ab.
* Has a history of complications of immunosuppression
* Suspected clinically relevant active hepatitis, including viral hepatitis, according to the investigator's judgment
* Known human immunodeficiency virus (HIV) infection
* Has a history of a diagnosis or condition that, in the judgment of the investigator, may affect study endpoint assessment or compromise participant safety.
* Received any non-study vaccine within 28 days before or after any dose of vaccine (except for seasonal influenza vaccine, which is not permitted within 14 days before or after any dose of vaccine)
* Received intravenous blood products (red blood cells, platelets, immunoglobulins) within 3 months prior to Day 1.
* Participated in an interventional clinical study within 28 days prior to Day 0 or plans to donate blood products while participating in this study.

Healthy Participants

Key Inclusion Criteria for Part A:

* In good general health without current or previous diagnosis of immunocompromising condition, immune-mediated disease, or other immunosuppressive condition, according to investigator assessment, at the time of consent, and has not been vaccinated with any COVID-19 vaccine at the time of consent.
* Understands, agrees, and is able to comply with the study procedures and provides written informed consent.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection (Day 1), agreement to continue adequate contraception or abstinence through 3 months following the second injection (Day 29), and not currently breastfeeding.
* Is medically stable, according to investigator's judgment, during the 3 months before signing consent.

Key Exclusion Criteria for Part A:

* Has a known close contact with anyone with laboratory confirmed SARS-CoV-2 infection or COVID-19 within 2 weeks prior to vaccine administration or known history of SARS-CoV-2 infection or positive SARS-CoV-2 test.
* Has prior or planned administration of a coronavirus vaccine (for example, SARS-CoV-2, SARS-CoV, or MERS-CoV vaccine).
* Has current treatment with investigational agents for either prophylaxis against COVID-19 or treatment of COVID-19 (for example, anti-SARS-CoV-2 monoclonal antibodies).
* Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation or that could interfere with safety assessments or interpretation of results according to the investigator's judgment.
* Has a history of a diagnosis or condition that, in the judgment of the investigator, may affect study endpoint assessment or compromise participant safety.
* Received any non-study vaccine within 28 days before or after any dose of vaccine (except for seasonal influenza vaccine, which is not permitted within 14 days before or after any dose of vaccine)
* Received intravenous blood products (red blood cells, platelets, immunoglobulins) within 3 months prior to Day 1.
* Received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids ≥20 mg/day of prednisone equivalent).
* Participated in an interventional clinical study within 28 days prior to Day 0 or plans to donate blood products while participating in this study.

Inclusion Criteria for Part B:

* Participants must have been previously enrolled in this study (mRNA-1273-P304), are actively participating in Part A, and at least 4 months from the last dose; or participant is either a kidney or a liver SOT recipient who is at least 90 days after transplantation at the time of consent and who completed primary vaccination series (3 doses for mRNA COVID-19 vaccine; 2 doses for non-mRNA COVID-19 vaccine or at least 1 dose of non-mRNA combined with 1 dose of mRNA COVID-19 vaccine) under the EUA who are at least 4 months from the last dose. All primary COVID-19 vaccination series must be completed after transplant.
* Female participants of childbearing potential may be enrolled in the study if the participant has a negative pregnancy test on the day of the first injection (booster dose Day 1).

Exclusion Criteria for Part B:

* Exclusion Criteria in Part A will apply except:

  1. prior or planned administration of a coronavirus vaccine and current treatment with investigational agents for either prophylaxis against COVID-19.
  2. known close contact with anyone with laboratory-confirmed SARS-CoV-2 infection or COVID-19 within 2 weeks prior to vaccine administration or any known history of SARS-CoV-2 infection or positive SARSCoV-2 test will apply only to new SOT participants who will be enrolled in Part B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Aventiv Research Inc, Mesa, Arizona
  - California Institute of Renal Research, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Tampa General Medical Group, Tampa, Florida
  - Piedmont Transplant Institute, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Northwell Health, Manhasset, New York
  - Colombia University Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Hospital, Cleveland, Ohio
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girard B, Figueroa AL, De Rosa SC, McElrath MJ, Azzi JR, Stolman D, Siangphoe U, de Windt E, Miller JM, Das R, Priddy F. mRNA-1273 COVID-19 vaccine induces CD4+ T-cell responses among solid organ transplant recipients. Front Immunol. 2025 Apr 3;16:1505871. doi: 10.3389/fimmu.2025.1505871. eCollection 2025. PMID 40248714
- [Derived] Figueroa AL, Azzi JR, Eghtesad B, Priddy F, Stolman D, Siangphoe U, Leony Lasso I, de Windt E, Girard B, Zhou H, Miller JM, Das R. Safety and Immunogenicity of the mRNA-1273 Coronavirus Disease 2019 Vaccine in Solid Organ Transplant Recipients. J Infect Dis. 2024 Sep 23;230(3):e591-e600. doi: 10.1093/infdis/jiae140. PMID 38513368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 214 solid organ transplant (SOT) participants (137 SOT kidney and 77 SOT liver participants) and 20 healthy participants were enrolled for the study.
Pre-assignment Details: Healthy participants cohort was included as a control group in the evaluation of humoral and cell-mediated immune response only; no comparisons of safety data with the healthy participants were made.
  Data reported for each arm in the Outcome Measures as specified in the Outcome Measure title.
Groups:
- Part A (Primary Series): Cohort A1 - SOT Participants: Unvaccinated SOT participants received 2 100-micrograms (μg) doses of mRNA-1273 vaccine by intramuscular (IM) injection, 28 days apart (on Day 1 and Day 29).
- Part A (Primary Series): Cohort A2 - SOT Participants: Unvaccinated SOT participants received 3 100-μg doses of mRNA-1273 vaccine by IM injection, on Day 1 and Day 29 (28 days apart) and on Day 85 (56 days after Dose 2).
- Part A (Primary Series): Cohort A3 - SOT Participants: Previously vaccinated SOT participants with 2 doses of Moderna COVID-19 vaccine outside the study received a single 100-μg dose (Dose 3) on Day 1.
- Part A (Primary Series): Cohort A5 - Healthy Participants: Healthy participants received 2 100-μg doses of mRNA-1273 vaccine by IM injection, 28 days apart (on Day 1 and Day 29).
- Part B (Booster Dose): Cohort B2 - SOT Participants: Unvaccinated SOT participants who received 3 doses of mRNA-1273 vaccine in Part A (Days 1, 29, and 85), received a 100-μg booster dose (BD) of mRNA-1273 vaccine on BD DAY 1.
- Part B (Booster Dose): Cohort B3 - SOT Participants: Previously vaccinated SOT participants with 2 doses of Moderna COVID-19 vaccine outside the study who received a single 100-μg dose (Dose 3) on Day 1 in Part A, received a 100-μg BD of mRNA-1273 vaccine on BD Day 1.
- Part B (Booster Dose): Cohort B4 - SOT Participants: SOT participants who completed primary vaccination with an mRNA or non-mRNA- COVID-19 vaccine outside mRNA-1273-P304, received a 100-μg BD of mRNA-1273 vaccine on BD Day 1.
- Part B (Booster Dose): Cohort B5 - Healthy Participants: Healthy participants who received 2 doses of mRNA-1273 vaccine in Part A (Days 1 and 29), received a 100-μg BD of mRNA-1273 vaccine on BD Day 1.
Period: Part A (Primary Series)
Arm/Group | Part A (Primary Series): Cohort A1 - SOT Participants | Part A (Primary Series): Cohort A2 - SOT Participants | Part A (Primary Series): Cohort A3 - SOT Participants | Part A (Primary Series): Cohort A5 - Healthy Participants | Part B (Booster Dose): Cohort B2 - SOT Participants | Part B (Booster Dose): Cohort B3 - SOT Participants | Part B (Booster Dose): Cohort B4 - SOT Participants | Part B (Booster Dose): Cohort B5 - Healthy Participants
Started | 3 | 58 | 71 | 20 | 0 | 0 | 0 | 0
Received First Study Injection | 3 | 58 | 0 | 20 | 0 | 0 | 0 | 0
Received Second Study Injection | 3 | 58 | 0 | 0 | 0 | 0 | 0 | 0
Received Third Study Injection | 0 | 57 | 71 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 57 | 71 | 17 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Part B (Booster Dose)
Arm/Group | Part A (Primary Series): Cohort A1 - SOT Participants | Part A (Primary Series): Cohort A2 - SOT Participants | Part A (Primary Series): Cohort A3 - SOT Participants | Part A (Primary Series): Cohort A5 - Healthy Participants | Part B (Booster Dose): Cohort B2 - SOT Participants | Part B (Booster Dose): Cohort B3 - SOT Participants | Part B (Booster Dose): Cohort B4 - SOT Participants | Part B (Booster Dose): Cohort B5 - Healthy Participants
Started | 0 | 0 | 0 | 0 | 33 | 44 | 82 | 10
Received Booster Injection | 0 | 0 | 0 | 0 | 33 | 44 | 81 | 10
Completed | 0 | 0 | 0 | 0 | 29 | 34 | 78 | 7
Not Completed | 0 | 0 | 0 | 0 | 4 | 10 | 4 | 3
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other Than Specified | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3 | 5 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Groups:
- SOT Kidney Participants: Unvaccinated or previously vaccinated SOT kidney participants received up to 3 100-μg doses of mRNA-1273 vaccine in Part A and a single 100-μg BD of mRNA-1273 vaccine in Part B.
- SOT Liver Participants: Unvaccinated or previously vaccinated SOT liver participants received up to 3 100-μg doses of mRNA-1273 vaccine in Part A and a single 100-μg BD of mRNA-1273 vaccine in Part B.
- Healthy Participants: Healthy participants received 2 doses of mRNA-1273 vaccine in Part A and a single 100-μg BD of mRNA-1273 vaccine in Part B.
- Total: Total of all reporting groups
Arm/Group | SOT Kidney Participants | SOT Liver Participants | Healthy Participants | Total
Number analyzed (Participants) | 137 | 77 | 20 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 108 | 58 | 18 | 184
  >=65 years | 29 | 19 | 2 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 38 | 10 | 110
  Male | 75 | 39 | 10 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 5 | 2 | 22
  Not Hispanic or Latino | 121 | 71 | 18 | 210
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 8 | 3 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 13 | 3 | 39
  White | 94 | 55 | 11 | 160
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 10 | 4 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Parts A and B: Number of SOT Participants With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was any AE reported by the participant that was not specified as a solicited adverse reaction (AR) or was specified as a solicited AR but started outside the protocol-defined period for reporting solicited ARs (that is, for the 7 days after each dose of vaccine). A summary of serious adverse events (SAEs) and all nonserious AEs ("Other") reported up to the end of the study (up to Day 419), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to 28 days post-vaccination
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Groups:
- SOT Total: Unvaccinated or previously vaccinated SOT kidney and liver participants received up to 3 100-μg doses of mRNA-1273 vaccine in Part A and a single 100-μg BD of mRNA-1273 vaccine in Part B.
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 137 | 77 | 214
Participants | 48 | 41 | 89

2. Primary Outcome: Parts A and B: Number of Healthy Participants With Unsolicited AEs
Description: An unsolicited AE was any AE reported by the participant that was not specified as a solicited AR or was specified as a solicited AR but started outside the protocol-defined period for reporting solicited ARs (that is, for the 7 days after each dose of vaccine). A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study (up to Day 419), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Up to 28 days post-vaccination
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 20
Participants | 12

3. Primary Outcome: Parts A and B: Number of SOT Participants With Medically-Attended Adverse Events (MAAEs)
Description: An MAAE was an AE that led to an unscheduled visit to an healthcare practitioner (HCP). This included visits to a study site for unscheduled assessments (for example, abnormal laboratory test results follow-up, COVID-19) and visits to HCPs external to the study site (for example, urgent care, primary care physician). MAAEs were also required by protocol for routine surveillance of participants with symptoms for COVID-19 infection (fever, shortness of breath, cough, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, and diarrhea). All confirmed symptomatic COVID-19 cases were recorded as MAAEs. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Throughout the study period (up to Day 450)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 137 | 77 | 214
Participants | 86 | 56 | 142

4. Primary Outcome: Parts A and B: Number of Healthy Participants With MAAEs
Description: An MAAE was an AE that led to an unscheduled visit to an HCP. This included visits to a study site for unscheduled assessments (for example, abnormal laboratory test results follow-up, COVID-19) and visits to HCPs external to the study site (for example, urgent care, primary care physician). MAAEs were also required by protocol for routine surveillance of participants with symptoms for COVID-19 infection (fever, shortness of breath, cough, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, and diarrhea). All confirmed symptomatic COVID-19 cases were recorded as MAAEs. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Throughout the study period (up to Day 394)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 20
Participants | 14

5. Primary Outcome: Parts A and B: Number of SOT Participants With Serious Adverse Events (SAEs)
Description: An AE (including an AR) was considered an SAE if, in the view of either the investigator or Sponsor, it results in any of the following outcomes: death, was life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly or birth defect, or medically important event. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Throughout the study period (up to Day 450)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 137 | 77 | 214
Participants | 29 | 19 | 48

6. Primary Outcome: Parts A and B: Number of Healthy Participants With SAEs
Description: as for outcome 5
Time Frame: Throughout the study period (up to Day 394)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 20
Participants | 1

7. Primary Outcome: Parts A and B: Number of SOT Participants With Adverse Event of Special Interests (AESIs), Including Myocarditis/Pericarditis
Description: An AESI was an AE (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Throughout the study period (up to Day 450)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 137 | 77 | 214
Participants | 15 | 13 | 28

8. Primary Outcome: Parts A and B: Number of Healthy Participants With AESIs, Including Myocarditis/Pericarditis
Description: as for outcome 7
Time Frame: Throughout the study period (up to Day 394)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 20
Participants | 1

9. Primary Outcome: Parts A and B: Number of SOT Participants With AEs Leading to Discontinuation From Dosing and/or Study Participation (Withdrawal)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug-related. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Throughout the study period (up to Day 450)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 137 | 77 | 214
Participants | 4 | 0 | 4

10. Primary Outcome: Parts A and B: Number of Healthy Participants With AEs Leading to Discontinuation From Dosing and/or Study Participation (Withdrawal)
Description: as for outcome 9
Time Frame: Throughout the study period (up to Day 394)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 20
Participants | 0

11. Primary Outcome: Parts A and B: Number of SOT Participants With Adjudicated Biopsy-Proven Organ Rejection
Description: A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Throughout the study period (up to Day 450)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 137 | 77 | 214
Participants | 1 | 2 | 3

12. Primary Outcome: Parts A and B: Number of Healthy Participants With Biopsy-Proven Organ Rejection
Description: as for outcome 11
Time Frame: Throughout the study period (up to Day 394)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 20
Participants | 0

13. Primary Outcome: Parts A and B: Number of SOT Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs, including local and systemic ARs were collected in the eDiary. Local ARs included: pain at injection site, erythema (redness) at injection site, swelling/induration (hardness) at injection site, and localized axillary swelling or tenderness ipsilateral to the injection arm. Systemic ARs included: headache, fatigue, myalgia (muscle aches all over the body), arthralgia (aching in several joints), nausea/vomiting, rash, body temperature (potentially fever), and chills. All solicited ARs (local and systemic) considered causally related to injection. ARs were graded 0-4 as reviewed and confirmed by Investigator; lower score indicates lower severity and a higher score indicates greater severity. Note, not all solicited ARs were considered AEs. The Investigator reviewed whether the solicited AR was also to be recorded as an AE. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 7 days post-vaccination
Population: Any study injection solicited safety set included all participants who received any (first, second, third, or booster) study injection and contributed any solicited AR data following that injection. Here, 'Number analyzed' signifies participants evaluable for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 137 | 77 | 214
Participants
  Solicited Local ARs: number analyzed (Participants) | 137 | 76 | 213
  Solicited Local ARs | 116 | 65 | 181
  Solicited Systemic ARs | 102 | 70 | 172

14. Primary Outcome: Parts A and B: Number of Healthy Participants With Solicited Local and Systemic ARs
Description: as for outcome 13
Time Frame: 7 days post-vaccination
Population: Any study injection solicited safety set included all participants who received any (first, second, third, or booster) study injection and contributed any solicited AR data following that injection.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 20
Participants
  Solicited Local ARs | 16
  Solicited Systemic ARs | 19

15. Primary Outcome: Part A: Geometric Mean Concentration (GMC) of Serum SARS-CoV-2-Specific Neutralizing Antibody (nAb) After the Second Dose in Unvaccinated Participants
Description: The GMC of VAC62 antibodies, as measured by pseudovirus neutralization assay (PsVNA) specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the lower limit of quantification (LLOQ) were replaced by 0.5*LLOQ. Values that were greater than the upper limit of quantification (ULOQ) were converted to the ULOQ if actual values were not available. LLOQ was 10 and ULOQ was 111433 arbitrary units (AU)/milliliter (mL). The 95% confidence intervals (CIs) were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GMC value, then back transformed to the original scale for presentation. Results in healthy participants were included as reference not for any comparisons.
Time Frame: Day 57 (for unvaccinated participants)
Population: The per protocol (PP) immunogenicity set (Part A) included all participants who received at least 1 dose of study drug, had no immunologic/virologic evidence of prior COVID-19 at baseline/pre-vaccination, had post-injection results available for at least 1 assay component corresponding to the immunogenicity analysis objective, and had no major protocol deviations that impacted immune response. 'Overall number of participants analyzed' = participants analyzed for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Groups:
- Part A: SOT Kidney (Unvaccinated Participants): Unvaccinated SOT kidney participants received up to 3 100-μg doses of mRNA-1273 vaccine in Part A.
- Part A: SOT Liver (Unvaccinated Participants): Unvaccinated SOT liver participants received up to 3 100-μg doses of mRNA-1273 vaccine in Part A.
- Healthy Participants: Healthy participants received 2 doses of mRNA-1273 vaccine in Part A.
Arm/Group | Part A: SOT Kidney (Unvaccinated Participants) | Part A: SOT Liver (Unvaccinated Participants) | Healthy Participants
Number analyzed (Participants) | 23 | 13 | 16
AU/mL | 54.2 [23.4 to 125.5] | 187.9 [67.6 to 522.6] | 1658.4 [951.1 to 2891.6]

16. Primary Outcome: Part A: GMC of SARS-CoV-2-Specific nAb 28 Days After Dose 3
Description: The GMC of VAC62 antibodies, as measured by PsVNA specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were converted to the ULOQ if actual values were not available. LLOQ was 10 and ULOQ was 111433 AU/mL. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GMC value, then back transformed to the original scale for presentation.
Time Frame: 28 days after Dose 3
Population: The PP immunogenicity set (Part A) included all participants who received at least 1 dose of study drug, had no immunologic/virologic evidence of prior COVID-19 at baseline/pre-vaccination, had post-injection results available for at least 1 assay component corresponding to the immunogenicity analysis objective, and had no major protocol deviations that impacted immune response. 'Overall number of participants analyzed' = participants analyzed for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Groups:
- SOT Kidney Participants: Unvaccinated or previously vaccinated SOT kidney participants received up to 3 100-μg doses of mRNA-1273 vaccine in Part A.
- SOT Liver Participants: Unvaccinated or previously vaccinated SOT liver participants received up to 3 100-μg doses of mRNA-1273 vaccine in Part A.
- SOT Total: Unvaccinated or previously vaccinated SOT kidney and liver participants received up to 3 100-μg doses of mRNA-1273 vaccine in Part A.
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 52 | 24 | 76
AU/mL | 353.5 [171.2 to 729.7] | 1340.2 [617.4 to 2909.1] | 538.4 [307.2 to 943.7]

17. Primary Outcome: Part B: GMC of SARS-CoV-2-Specific nAb 28 Days After the BD in SOT Participants Who Received the Moderna Primary Series and Non-Moderna Primary Series
Description: as for outcome 16
Time Frame: 28 days after BD injection (BD-Day 29)
Population: The PP set (Part B) included all participants who received BD of study drug, had no immunologic or virologic evidence of prior COVID-19 at pre-booster before the BD, had post-booster results available for at least 1 assay component corresponding to the immunogenicity analysis objective, and had no major protocol deviations that impacted immune response during the period corresponding to the immunogenicity analysis objective.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Groups:
- Part B: SOT Kidney Participants: SOT kidney participants who received Moderna and non-Moderna primary series vaccine and a single 100-μg BD of mRNA-1273 vaccine.
- Part B: SOT Liver Participants: SOT liver participants who received Moderna and non-Moderna primary series vaccine and a single 100-μg BD of mRNA-1273 vaccine.
Arm/Group | Part B: SOT Kidney Participants | Part B: SOT Liver Participants
Number analyzed (Participants) | 62 | 31
AU/mL | 430.7 [216.4 to 857.5] | 3946.0 [1944.5 to 8007.8]

18. Secondary Outcome: Part A: GMC of SARS-CoV-2-Specific nAb for Unvaccinated Participants Receiving the 2-Dose Regimen
Description: The GMC of VAC62 antibodies, as measured by pseudovirus neutralization assay PsVNA specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 10 and ULOQ was 111433 AU/mL. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GMC value, then back transformed to the original scale for presentation. Results in healthy participants were included as reference not for any comparisons. 95% CI cannot be calculated with an 'N' less than 2.
Time Frame: Days 1, 28 days after Dose 1, 28 days after Dose 2, 6 months after Dose 2, and 1 year after Dose 2
Population: PP immunogenicity set (Part A): all participants who received at least 1 dose of study drug, had no immunologic/virologic evidence of prior COVID-19 at baseline, had post-injection results available for at least 1 assay component corresponding to immunogenicity analysis, and had no major protocol deviations that impacted immune response. 'Overall number of participants analyzed' = participants analyzed for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part A: SOT Kidney (Unvaccinated Participants) | Part A: SOT Liver (Unvaccinated Participants) | Healthy Participants
Number analyzed (Participants) | 24 | 14 | 16
AU/mL
  Day 1 | 13.9 [10.1 to 19.2] | 13.6 [8.0 to 23.2] | 11.2 [7.3 to 17.1]
  28 days after Dose 1: number analyzed (Participants) | 22 | 14 | 16
  28 days after Dose 1 | 18.6 [11.1 to 31.2] | 28.4 [15.2 to 53.1] | 58.2 [31.4 to 107.8]
  28 days after Dose 2: number analyzed (Participants) | 23 | 13 | 16
  28 days after Dose 2 | 54.2 [23.4 to 125.5] | 187.9 [67.6 to 522.6] | 1658.4 [951.1 to 2891.6]
  6 months after Dose 2: number analyzed (Participants) | 1 | 1 | 14
  6 months after Dose 2 | 859.0 | 4134.0 | 948.5 [322.7 to 2787.6]
  1 year after Dose 2: number analyzed (Participants) | 1 | 1 | 4
  1 year after Dose 2 | 412.0 | 7285.0 | 1439.3 [100.8 to 20561.0]

19. Secondary Outcome: Part A: GMC of SARS-CoV-2-Specific nAb for Unvaccinated and Previously Vaccinated Participants Receiving the 3-Dose Regimen
Description: The GMC of VAC62 antibodies, as measured by pseudovirus neutralization assay PsVNA specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 10 and ULOQ was 111433 AU/mL. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GMC value, then back transformed to the original scale for presentation. Results in healthy participants were included as reference not for any comparisons.
Time Frame: 28 days after Dose 3, 6 months after Dose 3, and 1 year after Dose 3
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 52 | 24 | 76
AU/mL
  28 days after Dose 3 | 353.5 [171.2 to 729.7] | 1340.2 [617.4 to 2909.1] | 538.4 [307.2 to 943.7]
  6 months after Dose 3: number analyzed (Participants) | 24 | 6 | 30
  6 months after Dose 3 | 222.5 [72.7 to 681.4] | 867.2 [62.9 to 11960.3] | 292.1 [109.1 to 782.0]
  1 year after Dose 3: number analyzed (Participants) | 13 | 2 | 15
  1 year after Dose 3 | 990.7 [198.6 to 4942.3] | 480.8 [NA to 4400000000000] — Result below the LLOQ. | 899.7 [217.0 to 3729.4]

20. Secondary Outcome: Part A: GMFR of nAb for Unvaccinated Participants Receiving the 2-Dose Regimen Relative to Day 1
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. The GMFR of VAC62 antibodies, as measured by PsVNA specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 10 and ULOQ was 111433 AU/mL. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GMC value, then back transformed to the original scale for presentation. Results in healthy participants were included as reference not for any comparisons. 95% CI cannot be calculated with an 'N' less than 2.
Time Frame: 28 days after Dose 1, 28 days after Dose 2, 6 months after Dose 2, and 1 year after Dose 2
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part A: SOT Kidney (Unvaccinated Participants) | Part A: SOT Liver (Unvaccinated Participants) | Healthy Participants
Number analyzed (Participants) | 23 | 14 | 16
ratio
  28 days after Dose 1 | 1.3 [0.8 to 2.1] | 2.1 [0.9 to 5.0] | 5.2 [2.7 to 9.9]
  28 days after Dose 2: number analyzed (Participants) | 23 | 13 | 16
  28 days after Dose 2 | 3.7 [1.7 to 8.2] | 13.8 [3.7 to 51.9] | 148.4 [84.3 to 261.2]
  6 months after Dose 2: number analyzed (Participants) | 1 | 1 | 14
  6 months after Dose 2 | 171.8 | 826.8 | 96.4 [36.8 to 252.8]
  1 year after Dose 2: number analyzed (Participants) | 1 | 1 | 4
  1 year after Dose 2 | 82.4 | 1457.0 | 145.1 [11.8 to 1778.7]

21. Secondary Outcome: Part A: GMFR of nAb for Unvaccinated and Previously Vaccinated Participants Receiving the 3-Dose Regimen Relative to Day 1
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. The GMFR of VAC62 antibodies, as measured by PsVNA specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 10 and ULOQ was 111433 AU/mL. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GMC value, then back transformed to the original scale for presentation. Results in healthy participants were included as reference not for any comparisons.
Time Frame: 28 days after Dose 3, 6 months after Dose 3, 1 year after Dose 3
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 22 | 11 | 33
ratio
  28 days after Dose 3 | 16.6 [6.6 to 41.7] | 56.8 [10.5 to 306.4] | 25.0 [11.2 to 55.9]
  6 months after Dose 3: number analyzed (Participants) | 12 | 6 | 18
  6 months after Dose 3 | 16.2 [4.2 to 62.7] | 65.8 [3.0 to 1429.9] | 25.8 [7.7 to 86.7]
  1 year after Dose 3: number analyzed (Participants) | 13 | 2 | 15
  1 year after Dose 3 | 990.7 [198.6 to 4942.3] | 480.8 [NA to 4400000000000] — Result below the LLOQ. | 899.7 [217.0 to 3729.4]

22. Secondary Outcome: Part A: Geometric Mean (GM) Value of Anti-SARS-CoV-2 S-specific Binding Antibody (bAb) for Unvaccinated Participants Receiving the 2-Dose Regimen
Description: The GM level of VAC123 spike antibodies, as measured by MesoScale Discovery (MSD) electrochemiluminescence (ECL) multiplex assay specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 69 and ULOQ was 14400000 AU/mL. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GM value, then back transformed to the original scale for presentation. Results in healthy participants were included as reference not for any comparisons. 95% CI cannot be calculated with an 'N' less than 2.
Time Frame: Days 1, 28 days after Dose 1, 28 days after Dose 2, 6 months after Dose 2, and 1 year after Dose 2
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part A: SOT Kidney (Unvaccinated Participants) | Part A: SOT Liver (Unvaccinated Participants) | Healthy Participants
Number analyzed (Participants) | 24 | 14 | 16
AU/mL
  Day 1 | 68.3 [39.9 to 116.9] | 59.1 [33.6 to 104.0] | 53.6 [34.4 to 83.4]
  28 days after Dose 1: number analyzed (Participants) | 23 | 14 | 16
  28 days after Dose 1 | 346.4 [127.7 to 939.6] | 1213.9 [269.5 to 5467.4] | 23668.2 [13462.8 to 41609.8]
  28 days after Dose 2: number analyzed (Participants) | 23 | 13 | 16
  28 days after Dose 2 | 3190.1 [828.4 to 12284.7] | 20734.0 [3689.2 to 116527.2] | 272797.7 [188489.1 to 394816.2]
  6 months after Dose 2: number analyzed (Participants) | 1 | 1 | 14
  6 months after Dose 2 | 84460.0 | 202997.0 | 97534.9 [47881.0 to 198681.0]
  1 year after Dose 2: number analyzed (Participants) | 1 | 1 | 4
  1 year after Dose 2 | 44828.0 | 167863.0 | 161241.8 [19006.2 to 1367917.7]

23. Secondary Outcome: Part A: GM Value of Anti-SARS-CoV-2 S-specific bAb for Unvaccinated and Previously Vaccinated Participants Receiving the 3-Dose Regimen
Description: The GM level of VAC123 spike antibodies, as measured by MSD ECL multiplex assay specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 69 and ULOQ was 14400000 AU/mL. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GM value, then back transformed to the original scale for presentation. Results in healthy participants were included as reference not for any comparisons.
Time Frame: 28 days after Dose 3, 6 months after Dose 3, and 1 year after Dose 3
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 53 | 24 | 77
AU/mL
  28 days after Dose 3 | 26674.0 [10865.9 to 65480.5] | 167141.1 [69651.7 to 401083.3] | 47260.9 [23657.2 to 94415.1]
  6 months after Dose 3: number analyzed (Participants) | 24 | 6 | 30
  6 months after Dose 3 | 19289.6 [5878.6 to 63295.3] | 69076.5 [12838.6 to 371658.0] | 24895.7 [9274.4 to 66828.7]
  1 year after Dose 3: number analyzed (Participants) | 13 | 2 | 15
  1 year after Dose 3 | 66847.7 [16994.7 to 262942.2] | 42266.8 [NA to 664919284614.9] — Result below the LLOQ. | 62884.2 [18998.9 to 208139.7]

24. Secondary Outcome: Part A: Geometric Mean Fold-Rise (GMFR) of bAb for Unvaccinated Participants Receiving the 2-Dose Regimen Relative to Day 1
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. The GMFR of VAC123 spike antibodies, as measured by MSD ECL multiplex assay specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 69 and ULOQ was 14400000 AU/mL. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GMFR, then back transformed to the original scale for presentation. Results in healthy participants were included as reference not for any comparisons. 95% CI cannot be calculated with an 'N' less than 2.
Time Frame: 28 days after Dose 1, 28 days after Dose 2, 6 months after Dose 2, and 1 year after Dose 2
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part A: SOT Kidney (Unvaccinated Participants) | Part A: SOT Liver (Unvaccinated Participants) | Healthy Participants
Number analyzed (Participants) | 23 | 14 | 16
ratio
  28 days after Dose 1 | 4.9 [1.8 to 13.4] | 20.5 [4.3 to 97.0] | 441.9 [244.5 to 798.5]
  28 days after Dose 2: number analyzed (Participants) | 23 | 13 | 16
  28 days after Dose 2 | 45.4 [10.7 to 191.8] | 399.0 [64.0 to 2488.0] | 5092.9 [3032.6 to 8553.1]
  6 months after Dose 2: number analyzed (Participants) | 1 | 1 | 14
  6 months after Dose 2 | 2448.1 | 5884.0 | 1710.0 [755.9 to 3868.5]
  1 year after Dose 2: number analyzed (Participants) | 1 | 1 | 4
  1 year after Dose 2 | 1299.4 | 4865.6 | 2567.2 [47.8 to 137952.8]

25. Secondary Outcome: Part A: GMFR of bAb for Unvaccinated and Previously Vaccinated Participants Receiving the 3-Dose Regimen Relative to Day 1
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. The GMFR of VAC123 spike antibodies, as measured by MSD ECL multiplex assay specific to the SARS-CoV-2 spike protein is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ. Values that were greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 69 and ULOQ was 14400000 AU/mL. The 95% CIs were calculated based on the t-distribution of the log-transformed values or the difference in the log-transformed values for GMFR, then back transformed to the original scale for presentation. Results in healthy participants were included as reference not for any comparisons.
Time Frame: 28 days after Dose 3, 6 months after Dose 3, 1 year after Dose 3
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 22 | 11 | 33
ratio
  28 days after Dose 3 | 275.5 [60.9 to 1246.2] | 1556.2 [219.1 to 11051.0] | 490.7 [151.8 to 1586.4]
  6 months after Dose 3: number analyzed (Participants) | 12 | 6 | 18
  6 months after Dose 3 | 554.9 [161.0 to 1912.2] | 824.1 [124.9 to 5436.5] | 633.1 [251.7 to 1592.5]
  1 year after Dose 3: number analyzed (Participants) | 8 | 2 | 10
  1 year after Dose 3 | 690.8 [71.7 to 6656.9] | 746.2 [NA to 6400000000000] — Result below the LLOQ. 6400000000000 | 701.5 [114.3 to 4305.5]

26. Secondary Outcome: Part A: Number of SOT Participants With Asymptomatic SARS-CoV-2 Infection
Description: Asymptomatic SARS-CoV-2 infection was identified by absence of COVID-19 symptoms and infections as detected by reverse transcriptase polymerase chain reaction (RT-PCR) central or local test or serology test as binding antibody (bAb) level against SARS-CoV-2 nucleocapsid protein negative (as measured by Roche Elecsys) at Day 1 that became positive (as measured by Roche Elecsys) post-baseline or positive RT-PCR (CLIA-certified central or local) laboratory post-baseline at scheduled or unscheduled/illness visits. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study (up to Day 419), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 14 days after second and third injection
Population: The modified intent-to-treat (mITT) set (Part A) included all participants who received at least 1 dose of study drug, had no immunologic or virologic evidence of prior COVID-19 at baseline/pre-vaccination before the first dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A (Primary Series): Cohort A1 (SOT Kidney Participants): Unvaccinated SOT kidney participants received 2 100-μg doses of mRNA-1273 vaccine by IM injection, 28 days apart (on Day 1 and Day 29).
- Part A (Primary Series): Cohort A1 (SOT Liver Participants): Unvaccinated SOT liver participants received 2 100-μg doses of mRNA-1273 vaccine by IM injection, 28 days apart (on Day 1 and Day 29).
- Part A (Primary Series): Cohort A2 and A3 (SOT Kidney Participants): Unvaccinated or previously vaccinated SOT kidney participants received 2 100-μg doses of mRNA-1273 vaccine by IM injection, 28 days apart (on Day 1 and Day 29). Participants also receive a third dose (100-μg) of mRNA-1273 vaccine on Day 85 (56 days after Dose 2).
- Part A (Primary Series): Cohort A2 and A3 (SOT Liver Participants): Unvaccinated or previously vaccinated SOT liver participants received 2 100-μg doses of mRNA-1273 vaccine by IM injection, 28 days apart (on Day 1 and Day 29). Participants also receive a third dose (100-μg) of mRNA-1273 vaccine on Day 85 (56 days after Dose 2).
Arm/Group | Part A (Primary Series): Cohort A1 (SOT Kidney Participants) | Part A (Primary Series): Cohort A1 (SOT Liver Participants) | Part A (Primary Series): Cohort A2 and A3 (SOT Kidney Participants) | Part A (Primary Series): Cohort A2 and A3 (SOT Liver Participants)
Number analyzed (Participants) | 2 | 1 | 70 | 45
Participants | 0 | 1 | 8 | 4

27. Secondary Outcome: Part A: Number of Healthy Participants With Asymptomatic SARS-CoV-2 Infection
Description: Asymptomatic SARS-CoV-2 infection was identified by absence of COVID-19 symptoms and infections as detected by reverse transcriptase polymerase chain reaction (RT-PCR1) central or local test or serology test as bAb level against SARS-CoV-2 nucleocapsid protein negative (as measured by Roche Elecsys) at Day 1 that became positive (as measured by Roche Elecsys) post-baseline or positive RT-PCR (CLIA-certified central or local) laboratory post-baseline at scheduled or unscheduled/illness visits. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study (up to Day 419), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 14 days after second and third injection
Population: The mITT set (Part A) included all participants who received at least 1 dose of study drug, had no immunologic or virologic evidence of prior COVID-19 at baseline/pre-vaccination before the first dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 17
Participants | 4

28. Secondary Outcome: Part A: Number of SOT Participants With the Occurrence of COVID-19
Description: COVID-19 case was identified as a positive post-baseline RT-PCR (CLIA-certified central or local) laboratory for SARS-CoV-2, together with at least 2 systemic symptoms: fever (≥ 38 degree celsius [°C]/≥ 100.4 degree fahrenheit [°F]), chills, myalgia, headache, sore throat, new olfactory and taste disorder(s), or at least 1 of the following respiratory signs/symptoms: cough, shortness of breath or difficulty breathing, or clinical or radiographical evidence of pneumonia. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study (up to Day 419), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 14 days after second and third injection
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Primary Series): Cohort A1 (SOT Kidney Participants) | Part A (Primary Series): Cohort A1 (SOT Liver Participants) | Part A (Primary Series): Cohort A2 and A3 (SOT Kidney Participants) | Part A (Primary Series): Cohort A2 and A3 (SOT Liver Participants)
Number analyzed (Participants) | 2 | 1 | 70 | 45
Participants | 0 | 0 | 12 | 7

29. Secondary Outcome: Part A: Number of Healthy Participants With the Occurrence of COVID-19
Description: COVID-19 case was identified as a positive post-baseline RT-PCR (CLIA-certified central or local) laboratory for SARS-CoV-2, together with at least 2 systemic symptoms: fever (≥ 38°C/≥ 100.4°F), chills, myalgia, headache, sore throat, new olfactory and taste disorder(s), or at least 1 of the following respiratory signs/symptoms: cough, shortness of breath or difficulty breathing, or clinical or radiographical evidence of pneumonia. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study (up to Day 419), regardless of causality, is located in the Reported "Adverse Events" section. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study (up to Day 419), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 14 days after second and third injection
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 17
Participants | 2

30. Secondary Outcome: Part A: Number of SOT Participants With the Occurrence of Severe COVID-19
Description: Severe COVID-19 case was identified as a COVID-19 case (RT-PCR [CLIA-certified central or local] laboratory) for SARS-CoV-2, together with any of the following: respiratory rate ≥30 per minute, heart rate ≥125 beats per minute, oxygen saturation(SpO2) ≤93% on room air at sea level, or partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FIO2) <300 millimeters of mercury (mmHg); or respiratory failure or acute respiratory distress syndrome (ARDS), defined as needing high-flow oxygen, noninvasive or mechanical ventilation, or extracorporeal membrane oxygenation) or evidence of shock (systolic blood pressure <90 mm Hg, diastolic BP <60 mm Hg, or requiring vasopressors); or significant acute renal, hepatic, or neurologic dysfunction; OR admission to an intensive care unit or death. A summary of SAEs and all nonserious AEs ("Other") reported up to the end of the study (up to Day 419), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: 14 days after second and third injection
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Primary Series): Cohort A1 (SOT Kidney Participants) | Part A (Primary Series): Cohort A1 (SOT Liver Participants) | Part A (Primary Series): Cohort A2 and A3 (SOT Kidney Participants) | Part A (Primary Series): Cohort A2 and A3 (SOT Liver Participants)
Number analyzed (Participants) | 2 | 1 | 70 | 45
Participants | 0 | 0 | 1 | 2

31. Secondary Outcome: Part A: Number of Healthy Participants With the Occurrence of Severe COVID-19
Description: as for outcome 30
Time Frame: 14 days after second and third injection
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants
Number analyzed (Participants) | 17
Participants | 0

32. Secondary Outcome: Parts A and B: Number of SOT Participants Who Changed Immunosuppressant Therapy
Description: A summary of serious adverse events (SAEs) and all nonserious AEs ("Other") reported up to the end of the study (up to Day 419), regardless of causality, is located in the Reported "Adverse Events" section.
Time Frame: Throughout the study period (up to Day 450)
Population: Safety set included all participants who received at least 1 dose of study drug in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total
Number analyzed (Participants) | 137 | 77 | 214
Participants | 52 | 37 | 89

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events were collected throughout the entire period of the study (from Day 1 up to the end of study [Day 450]). Unsolicited AEs were collected for 28 days after the vaccination.
Description: The safety analysis population consisted of all randomized participants who received at least 1 dose of vaccine. Unsolicited AEs were evaluated via the electronic case report form (eCRF) by the investigator at each visit. Study participants may have experienced both serious and non-serious event during the study. Thus, the same event in the same participant is summarized in both Serious Adverse Events and Other (Not Including Serious) Adverse Events table.
Arm/Group | SOT Kidney Participants | SOT Liver Participants | SOT Total | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 4/137 | 0/77 | 4/214 | 0/20
Serious Adverse Events (participants affected / at risk) | 28/137 | 17/77 | 45/214 | 1/20
Other Adverse Events (participants affected / at risk) | 49/137 | 38/77 | 87/214 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOT Kidney Participants (N=137) | SOT Liver Participants (N=77) | SOT Total (N=214) | Healthy Participants (N=20)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis escherichia coli (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (6) | 0 (0) | 4 (6) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Liver transplant rejection (Immune system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (5) | 3 (6) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 1 (1) | 2 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 9 (13) | 2 (2) | 11 (15) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis meckel's (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOT Kidney Participants (N=137) | SOT Liver Participants (N=77) | SOT Total (N=214) | Healthy Participants (N=20)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 3 (4)
Rhinovirus infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (4) | 6 (7) | 0 (0)
Urinary tract infection (Infections and infestations) | 14 (19) | 5 (8) | 19 (27) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ageusia (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 0 (0) | 4 (5) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 5 (5) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 3 (3) | 10 (10) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 4 (4) | 7 (9) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 7 (7) | 1 (1)
Faecalith (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (6) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 5 (5) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 6 (6) | 8 (8) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 5 (6) | 6 (8) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 10 (11) | 7 (8) | 17 (19) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 3 (5) | 5 (7) | 0 (0)
Blood urea increased (Investigations) | 2 (2) | 4 (4) | 6 (6) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Superficial injury of eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Healthy participants cohort was included as a control group in the evaluation of humoral and cell-mediated immune response only; no comparisons of safety data with the healthy participants were made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT04860297/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT04860297/SAP_001.pdf